CLINICAL TRIAL: NCT06425328
Title: Effect of Nutritional Habits on Oral Microbiota in Adolescents
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Betül Cicek, Professor, TC Erciyes University
Other Study IDs: ErciyesU-BVD-BAG-01
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Nutrition, Healthy; Adolescent Behavior; Microbial Colonization
Keywords: adolescent; Nutritional Sciences; Oral Health
MeSH Terms: conditions — Adolescent Behavior; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Saliva samples were taken from all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Underweight: BMI calculation was calculated with the equation "body weight (kg) / height (m)2" using body weight and height measurement results. BMI was evaluated according to the World Health Organization's BMI Z score classification for ages 5-19. Accordingly, those with a BMI z score below -1 SD are defined as underweight.
- Normal weight: BMI calculation was calculated with the equation "body weight (kg) / height (m)2" using body weight and height measurement results. BMI was evaluated according to the World Health Organization's BMI Z score classification for ages 5-19. Accordingly, BMI z scores between -1 SD +1 SD are defined as normal weight.
- Overweight: BMI calculation was calculated with the equation "body weight (kg) / height (m)2" using body weight and height measurement results. BMI was evaluated according to the World Health Organization's BMI Z score classification for ages 5-19. Accordingly, those with a BMI z score between +1 SD +2 SD are defined as overweight
- Obese: BMI calculation was calculated with the equation "body weight (kg) / height (m)2" using body weight and height measurement results. BMI was evaluated according to the World Health Organization's BMI Z score classification for ages 5-19. Accordingly, those with a BMI z score above +2 SD are defined as obese.

SUMMARY:
The aim of this study is to examine the relationship between oral microbiota and eating habits, sleep quality and hedonic hunger in adolescents.

DETAILED DESCRIPTION:
Oral microbiota; While it is associated with systemic diseases such as obesity, diabetes and cancer, it is also associated with oral diseases such as oral cancers, tooth decay and gum diseases. Nutrition is seen as an important factor in maintaining oral health. In particular, the amount and frequency of sugar consumption, the type and consistency of food, the frequency of eating, the consumption of cariogenic foods with other foods and the duration of carbohydrates remaining on the teeth are among the factors that affect oral health. The aim of this study is to examine the relationship between oral microbiota and eating habits, sleep quality and hedonic hunger in adolescents. The study is planned to be carried out in 4 stages. First stage; A survey form will be filled out that questions general information about children, oral health practices, nutritional habits and frequency of food consumption. In the second stage; Children's anthropometric measurements (body weight (kg), height (cm), waist circumference (cm) will be taken and bioelectrical impedance analysis (BIA) results will be recorded. In the third stage, oral examinations of the children will be performed. In the final stage, saliva samples of the children will be collected. Bacteria Logarithmic values will be used when comparing the concentrations between groups. The suitability of the parameters to normal distribution will be evaluated with q-q graphs and Shapiro-Wilk test. Student t test will be used for variables that comply with normal distribution and Mann Whitney U test will be used for changes that do not comply with normal distribution. The relationship will be evaluated with the Spearman or Pearson correlation test according to the normality distribution. IBM SPSS (Statistical Package for Social Sciences) 22.0 package program will be used when evaluating the data obtained as a result of the study. While examining the hypothesis tests, α = 0.05 and accordingly the confidence interval will be determined as 95%. It will be evaluated at p<0.05 level. In order to enable healthy adolescents to reach a good standard of living, there is a need for a more accurate understanding of the relationship between oral microbiota, nutrition and sleep. As a result of this study, it is aimed to reveal the relationship between oral microbiota and eating habits, sleep quality and hedonic hunger in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* 14-16 years old
* Not receiving special medical nutrition therapy
* No chronic systemic disease, nutritional disorder and/or endocrine disease that may affect growth and development
* Adolescents without congenital developmental disorders

Exclusion Criteria:

* Those who had any severe oral disease or periodontal treatment including supragingival curettage and root planning before the study
* Those who used any antibiotic, anti-inflammatory or sedative medication until 3 months before the study
* Those with bleeding gums on the working day or within the previous 4 weeks
* Those who smoke

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study included 40 adolescents aged 14-16, who were thin, healthy, slightly overweight and obese, who applied to İsmet Yılmaz Akansu Family Health Center and met the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Oral microbiome characteristics | 1 month
  For oral microbiota analysis, saliva samples were taken from children who had brushed their teeth in the morning and had not consumed any food until 2 hours before, and microbiological procedures were performed. Saliva samples taken from all patients participating in the study were stored at -80°C until analysis. Saliva samples collected during the research process were transported to the center where the analyzes were carried out by preserving the cold chain, and DNA isolation and sequence analysis were carried out together with molecular biologists. DNA purification from saliva samples was carried out using standard commercial methods. In the polymerase chain reaction-based amplification of bacterial 16S rRNA sequences, primers belonging to the V3-V4 region, which were previously defined and stated to be suitable for the detection of bacterial diversity, were used.

SECONDARY OUTCOMES:
Anthropometric Measurements | 1 month
  BMI calculation was calculated with the equation "body weight (kg) / height (m)2" using body weight and height measurement results. BMI was evaluated according to the World Health Organization's BMI Z score classification for ages 5-19.
3 day food consumption record | 1 month
  On the first day of the food consumption record, a 24-hour retrospective was taken by the researcher, and on the other days, it was recorded in detail by telephone.
Oral Examination | 1 month
  Intraoral examination of all children in the study group was performed by sitting on a chair by the window and using a mirror-probe in daylight. Intraoral examination of all children was performed by a single pediatric dentist (E.D.) and recorded in the patient information form. The total number of decayed, missing and filled teeth (Decayed, Missing, And Filled Teeth: DMFT) and tooth surfaces (Decayed, Missing, And Filled Surfaces: DMFS) were calculated.
Pittsburg sleep quality index | 1 month
  It is a 19-question survey that evaluates sleep quality and disorders by scoring them over a one-month period. The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Children's Power of Food Scale | 1 month
  It is a 15-question survey developed to be used to determine hedonic hunger in school-age children. Items are rated on a 5-point Likert scale and summed to create a total score. Higher scores reflect greater responsiveness to the food environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No